CLINICAL TRIAL: NCT06571981
Title: Comparison Between Conventional Ultrasound and Remote Ultraportable ulTrasound for Abdominal Examination in the Context of Viral Hepatitis
Brief Title: Conventional Ultrasound Versus Remote Ultraportable ulTrasound in the Context of Viral Hepatitis
Acronym: RUTH
Status: Recruiting | Type: Observational
Sponsor: Naik Vietti Violi (Other)
Responsible Party: Sponsor-Investigator, Naik Vietti Violi, PD & MERc, Executive Physician of Diagnostic And Interventional Radiology Department, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Other Study IDs: BASEC 2024-D0048
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis; Teleradiology
MeSH Terms: conditions — Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with viral hepatitis: Every outpatient referred to the radiology department by a prescriber for abdominal US in the context of viral hepatitis
  Interventions: Device: TUP ultraportable US with teleradiology capacities; Device: CUS conventional ultrasound

INTERVENTIONS:
Device: TUP ultraportable US with teleradiology capacities — Comparison of abdominal ultrasound examinations in an at-risk population diagnosed with viral hepatitis: Ultraportable ultrasound with teleradiology capacities (TUP) versus conventional ultrasound (CUS).
Device: CUS conventional ultrasound — Comparison of abdominal ultrasound examinations in an at-risk population diagnosed with viral hepatitis: Ultraportable ultrasound with teleradiology capacities (TUP) versus conventional ultrasound (CUS).

SUMMARY:
Comparison of abdominal US exam in patients with viral hepatitis between ultraportable US with teleradiology capacities (TUP) versus conventional ultrasound (CUS)

DETAILED DESCRIPTION:
Primary Objective The investigation seeks primarily to determine the performance of abdominal US examinations realized with TUP and CUS based on defined imaging criteria Secondary Objectives Evaluate satisfaction and comfort and reproducibility of use of the ultraportable US

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* All adult patients with viral hepatitis for which an ultrasound is planned

Exclusion Criteria:

* Known or suspected non-compliance
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Previous enrollment into the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every outpatient referred to the radiology department by a prescriber for abdominal US in the context of viral hepatitis
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of TUP versus CUS for abdominal imaging in patients with viral hepatitis according to US LI-RADS categories ) for liver lesions | At the end of intervention
  LI RADS categories
  No observation OR Only definitely benign observation(s) Observation(s) < 10 mm in diameter, not definitely benign Observation(s) ≥ 10 mm in diameter, not definitely benign OR New thrombus in vein

SECONDARY OUTCOMES:
liver visualization scores | At the end of intervention
  no or minimal limitations; moderate limitations; severe limitations
liver surface nodularity | At the end of intervention
  Yes/No
focal lesions | At the end of intervention
  Yes/No
caudate lobe dimensions | At the end of intervention
  cm
portal flow velocity | At the end of intervention
  cm/s
biliary tract / gallbladder abnormalities | At the end of intervention
  Yes/No
lymph nodes presence | At the end of intervention
  Yes/No
free fluid | At the end of intervention
  Yes/No
examination time | At the end of intervention
  minutes
audio quality | At the end of intervention
  Adequate/Non Adequate
video quality | At the end of intervention
  Adequate/Non Adequate
patient's satisfaction | At the end of intervention
  Yes/No
agreement rates between reports | At the end of intervention
  Category 1: complete agreement/matching with teleradiologists reports; Category 2: minor discrepancy that would not impact patient management which included hedging terminology and ambiguous differences, for example fatty versus moderate fatty liver; Category 3: major discrepancy that would likely have an impact/change on patient management but would not lead to an adverse outcome for the patient; Category 4: major discrepancy that would impact patient management and lead to adverse outcomes for the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Naïk Vietti Violi, MD, Study Director — CHUV-UNIL
Locations (1):
- Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No